CLINICAL TRIAL: NCT04530214
Title: Predictive Elements of Trauma and Its After-effects: Importance of the Quality of Neurobiological Response to Stress
Acronym: LIFT-UP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2018PPRC30; 2019-A01811-56 (Other: IDRCB)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Stress Reaction
MeSH Terms: conditions — Fractures, Stress | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood collection — Blood collection at enrollment (before surgery) and at Visit 1 (45-60 days following surgery)
Other: Saliva collection — Saliva collection at enrollment (before surgery) and at Visit 1 (45-60 days following surgery)
Other: Electrocardiography (ECG) — Electrocardiography (ECG) at enrollment (24-72h following surgery) and at Visit 1 (45-60 days following surgery) to assess heart rate variability
Behavioral: Questionnaires — Mental health assessment through questionnaires at enrollment (24-72h following surgery), at Visit 1 (45-60 days following surgery), at Visit 2 (7 months following surgery) and at Visit 3 (12 months following surgery)

SUMMARY:
The neurobiological response to stress is an adaptive response allowing us to cope with the multiple aggressions of daily life. This response orchestrates the body's systemic reaction. The intensity of response to stress can modify the body's functioning, which implies a variety of fields where biomarkers may be isolated: immunity, psychology, neurophysiology, integrative physiology. When stress is too intense or prolonged, response to stress may become misfitted and deleterious.

This study is based on the hypothesis that a severe physical or psychological trauma is associated with an intense and misfitted stress that is responsible from an undue immuno-inflammatory activation (through sympathetic activation). The result is a subinvasive state of systemic and tissue inflammation (low-noise inflammation), responsible for the mid-term deleterious consequences of the traumatic event.

The objective of this study is to understand how the dysregulation of intense stress simultaneously generates an initial pathological state and an alteration of mid-term evolution (which is considered as a poor prognosis and/or as responsible for after-effects).

The investigators wish to identify relevant biomarkers of the mechanisms activated during intense stress and influencing the immuno-inflammatory and epigenetic spheres with deleterious consequences on physiological and psychological functions.

ELIGIBILITY:
Inclusion Criteria:

* Fracture of the upper end of the femur
* Cognitive state allowing the understanding of questionnaires

Exclusion Criteria:

* Traumatic Brain Injury
* Chronic inflammatory or immune pathologies
* On anticoagulants
* On neuroleptic or antidepressant treatment
* Pathology or health condition not allowing 1-year survival

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted to the emergency room for a fracture of the upper end of the femur.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of depression | 12 months following surgery
  Screening for depression will be done using a validated self-report questionnaire, the Geriatric Depression Scale Short Version (GDS).
  We will use the threshold value of 10 (score > or =) which corresponds to a very high probability of depression.
Occurrence of "psychosomatic death" | 12 months following surgery
  The diagnosis of "psychosomatic death" will be made by a physician. There is no consensus on the diagnosis of this syndrome. However, a patient with "psychosomatic death" is likely to be hospitalized or followed up medically and will not be able to respond to the investigator's request for a telephone interview.
Occurrence of death | 12 months following surgery
  Vital status will be collected from the participant's family or referring physician or at the birth & death record service (of the participant's town)

SECONDARY OUTCOMES:
Evolution of heart rate variability between enrollment and Visit 1 | Between enrollment and Visit 1 (45-60 days following surgery)
  Heart rate variability will be assessed using electrocardiography recordings
Evolution of perceived stress level between enrollment and Visit 1 | Between enrollment and Visit 1 (45-60 days following surgery)
  Perceived stress level will be assessed with the Perceived Stress Scale (PSS). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Evolution of anxiety level between enrollment and Visit 1 | Between enrollment and Visit 1 (45-60 days following surgery)
  Anxiety level will be assessed with the French version of Spielberger's State-Trait Anxiety Inventory adapted for people aged 65 and older (IASTA-Y65+).
  Individual scores on the IASTA-Y 65+ can range from 20 to 80 with higher scores indicating higher anxiety.
Evolution of post-traumatic stress disorder severity level between enrollment and Visit 1 | Between enrollment and Visit 1 (45-60 days following surgery)
  Post-traumatic stress disorder severity will be assessed with the Post-traumatic stress disorder CheckList for DSM-5 (Diagnostic and Statistical Manual Diploma in Social Medicine) (PCL-5) scale. Individual scores on the PCL-5 can range from 0 to 80 with higher scores indicating higher post-traumatic stress disorder severity.
Evolution of quality of life between enrollment and Visit 1 | Between enrollment and Visit 1 (45-60 days following surgery)
  Quality of life will be assessed using the abbreviated version of the World Health Organization Quality of Life (WHOQOL-Bref).
  The WHOQOL-Bref is grouped into 4 domains :
  * Physical health (score range from 7 to 35)
  * Psychological health (score range from 6 to 30)
  * Social relationships (score range from 3 to 15)
  * Environment (score range from 8-40) Higher scores indicate higher quality of life.
Evolution of cortisol level between enrollment and Visit 1 | Between enrollment and Visit 1 (45-60 days following surgery)
  Cortisol level will be measured in saliva sample.
Evolution of GABA level between enrollment and Visit 1 | Between enrollment and Visit 1 (45-60 days following surgery)
  Gamma-aminobutyric acid (GABA) level will be measured in blood sample.
Evolution of oxydative stress level between enrollment and Visit 1 | Between enrollment and Visit 1 (45-60 days following surgery)
  Oxydative stress level will be measured in blood sample.
Evolution of BDNF level between enrollment and Visit 1 | Between enrollment and Visit 1 (45-60 days following surgery)
  Brain-derived neurotrophic factor (BDNF) level will be measured in blood sample.
Evolution of pro and anti-inflammatory cytokines level between enrollment and Visit 1 | Between enrollment and Visit 1 (45-60 days following surgery)
  Cytokines level will be measured in blood sample.
Evolution of IGF-1 level between enrollment and Visit 1 | Between enrollment and Visit 1 (45-60 days following surgery)
  Insulin like growth factor type 1 (IGF-1) will be measured in blood sample.
Evolution of NPY level between enrollment and Visit 1 | Between enrollment and Visit 1 (45-60 days following surgery)
  Neuropeptide Y (NPY) level will be measured in blood sample.
Evolution of NPS between enrollment and Visit 1 | Between enrollment and Visit 1 (45-60 days following surgery)
  Neutrophil-platelet score (NPS) will be measured in blood sample.
Evolution of ocytocin level between enrollment and Visit 1 | Between enrollment and Visit 1 (45-60 days following surgery)
  Ocytocin level will be measured in blood sample.
Evolution of methylation of genes coding for BDNF between enrollment and Visit 1 | Between enrollment and Visit 1 (45-60 days following surgery)
  Methylation of genes coding for BDNF will be measured on DNA extracted from blood sample.
Evolution of methylation of genes coding for glucocorticoid receptors between enrollment and Visit 1 | Between enrollment and Visit 1 (45-60 days following surgery)
  Methylation of genes coding for glucocorticoid receptors will be measured on DNA extracted from blood sample.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Pellegrin, Bordeaux
  - Hôpital d'Instruction des Armées Percy, Clamart
  - Hôpital d'Instruction des Armées Bégin, Saint-Mandé
  - Hôpital d'Instruction des Armées Sainte-Anne, Toulon

IPD SHARING:
Plan to Share IPD: Undecided